CLINICAL TRIAL: NCT03313895
Title: Efficacy and Mechanisms of Combined Aerobic Exercise and Cognitive Training (ACT) in MCI
Brief Title: The Combined Aerobic Exercise and Cognitive Training (ACT) Trial: The ACT Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Rochester (Other); Mayo Clinic (Other); University of St Thomas (Unknown); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001135
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's disease; exercise; cognitive training; imaging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Motor Activity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cycling Only (Active Comparator): Moderate-intensity cycling, 3 times a week for 6 months, supervised by an exercise specialist
  Interventions: Behavioral: Cycling Only
- Cognitive Training Only (Active Comparator): Computerized cognitive training, 3 times a week for 6 months, supervised by a specialist
  Interventions: Behavioral: Cognitive Training Only
- ACT (Experimental): Moderate-intensity cycling followed by computerized cognitive training, 3 times a week for 6 months, supervised by a specialist
  Interventions: Behavioral: Aerobic & Cognitive Training (ACT)
- Stretching and Mental Stimulation Activities (Sham Comparator): Stretching and mental stimulation activities, 3 times a week for 6 months, supervised by a specialist
  Interventions: Behavioral: Stretching and Mental Stimulating Activities

INTERVENTIONS:
Behavioral: Aerobic & Cognitive Training (ACT) — ACT stands for combined aerobic exercise and cognitive training.
  Arms: ACT
Behavioral: Cycling Only — Cycling on a recumbent stationary cycle
  Arms: Cycling Only
Behavioral: Cognitive Training Only — Engage in cognitive training on a computer
  Arms: Cognitive Training Only
Behavioral: Stretching and Mental Stimulating Activities — Stretching exercises and mental stimulating activities on a computer
  Arms: Stretching and Mental Stimulation Activities

SUMMARY:
This multi-site clinical trial occurs at the University of Minnesota and University of Rochester. It tests the efficacy and additive/synergistic effects of an ACT intervention on cognition and relevant mechanisms (aerobic fitness, Alzheimer's disease [AD] signature cortical thickness, and default mode network [DMN]) in older adults with amnestic MCI (aMCI).

DETAILED DESCRIPTION:
Because almost all drug trials for Alzheimer's disease (AD) have failed, developing non-pharmacological interventions with strong potential to prevent or delay the onset of AD in high-risk populations (e.g., those with mild cognitive impairment [MCI]) is critically important. Aerobic exercise and cognitive training are 2 promising interventions for preventing AD. Aerobic exercise increases aerobic fitness, which in turn improves brain structure and function, while cognitive training improves selective neural function intensively. Hence, combined Aerobic exercise and Cognitive Training (ACT) may very well have an additive or synergistic effect on cognition by complementary strengthening of different neural functions. Few studies have tested ACT's effects, and those studies have reported discrepant findings, largely due to varying ACT programs. The purpose of this single-blinded, 2×2 factorial Phase II randomized controlled trial (RCT) is to test the efficacy and additive/synergistic effects of a 6-month combined cycling and speed of processing (SOP) training intervention on cognition and relevant mechanisms (aerobic fitness, AD signature cortical thickness, and functional connectivity in the default mode network [DMN]) in older adults with amnestic MCI (aMCI).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of MCI
* Community-dwelling
* Age 65 years and older
* English-speaking
* Adequate visual acuity
* Verified exercise safety by medical provider
* Stable on drugs affecting cognitive and psychological status
* Verified MRI safety
* Capacity to consent

Exclusion Criteria:

* Geriatric Depression Scale < 5
* Resting heart rate (HR) ≤50 due to arrhythmia or ≥100 beats/min
* Neurological (e.g., dementia, head trauma), psychiatric (e.g., bipolar, schizophrenia, or depression), or substance dependency (alcohol or chemical dependency) in the past 5 years that are the main contributor to MCI
* Contraindications to exercise, e.g. unstable angina, recent surgery
* New symptoms or diseases that have not been evaluated by a health care provider
* Current enrollment in another intervention study related to cognitive improvement (reduce confounding effects on outcomes)
* Abnormal MRI findings

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Executive function | Change from baseline to 3, 6, 12, and 18 months
  EXAMINER
Episodic memory | Change from baseline to 3, 6, 12, and 18 months
  RAVLT and BVMTR
AD-signature cortical thickness | Change from baseline to 6, 12, and 18 months
  Magnetic Resonance Imaging (MRI)
Functional connectivity in DMN | Change from baseline to 6, 12, and 18 months
  Functional MRI for Default Mode Network
Aerobic fitness | Change from baseline to 3, 6, 12, and 18 months
  VO2peak from symptom-limited peak cycle-ergometer test, and 10-m Incremental Shuttle Walk Test
Conversion to Alzheimer's disease | Change from baseline to 6, 12, and 18 months
  Clinical adjudication of Alzheimer's disease dementia

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yu, PhD, Principal Investigator — Arizona State University
Locations (4):
- United States (4):
  - Arizona State University, Phoenix, Arizona
  - Stanford University, Stanford, California
  - University of Minnesota, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derboghossian G, Pituch K, Anthony M, Salisbury D, Lin FV, Yu F. Relationships among cardiorespiratory fitness, brain age, and neurodegeneration in older adults with amnestic mild cognitive impairment. J Alzheimers Dis. 2025 Jun;105(3):945-954. doi: 10.1177/13872877251333613. Epub 2025 Apr 22. PMID 40262108
- [Derived] Salisbury DL, Lin FV, Yu F. Testing the iMplementation Framework fOr behavioral and LIfestyLe interventions in AlZheimer's DiseasE (MOBILIZE) via the ACT randomized controlled trial. Sci Rep. 2025 Feb 13;15(1):5341. doi: 10.1038/s41598-025-88890-9. PMID 39948366
- [Derived] Li D, Mielke MM, Bell WR, Reilly C, Zhang L, Lin FV, Yu F. Blood biomarkers as surrogate endpoints of treatment responses to aerobic exercise and cognitive training (ACT) in amnestic mild cognitive impairment: the blood biomarkers study protocol of a randomized controlled trial (the ACT Trial). Trials. 2020 Jan 6;21(1):19. doi: 10.1186/s13063-019-3798-1. PMID 31907024
- [Derived] Yu F, Lin FV, Salisbury DL, Shah KN, Chow L, Vock D, Nelson NW, Porsteinsson AP, Jack C Jr. Efficacy and mechanisms of combined aerobic exercise and cognitive training in mild cognitive impairment: study protocol of the ACT trial. Trials. 2018 Dec 22;19(1):700. doi: 10.1186/s13063-018-3054-0. PMID 30577848